CLINICAL TRIAL: NCT06893120
Title: Investigation of the Effectiveness of Cognitive Exercise Therapy Approach (BETY) in Parkinson's Disease
Brief Title: Cognitive Exercise Therapy Approach (BETY) in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Orkun Tüfekçi (Other)
Responsible Party: Sponsor-Investigator, Orkun Tüfekçi, Principal Investigator, PT, PhD(c), Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-06
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2022-09

CONDITIONS: Parkinson Disease
Keywords: Biopsychosocial model; depression; disease management; exercise; Parkinsons' Disease; quality of life
MeSH Terms: conditions — Parkinson Disease; Depression; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BETY session group (Experimental): Parkinson's Disease participating in BETY sessions.
  Interventions: Other: BETY
- Control Group (No Intervention): Control groups continued their disease management under the follow-up of their neurologists.

INTERVENTIONS:
Other: BETY — The cognitive Exercise Therapy Approach (Bilişsel Egzersiz Terapi Yaklaşımı-BETY) will be applied for 24 one-hour sessions, two days a week.
  Arms: BETY session group

SUMMARY:
Considering the impact of motor and non-motor findings on movement problems in the disease management of people living with PD, biopsychosocial evaluation and treatment approaches are essential. However, there are not many studies investigating the impact of a biopsychosocial-based exercise approach on the biopsychosocial characteristics of individuals in PD management.

The Cognitive Exercise Therapy Approach (BETY), an innovative exercise approach based on the biopsychosocial model, has been developed with the participation of individuals with rheumatism in exercise sessions for many years. This study investigated the effects of the BETY, a supervised biopsychosocial model-based exercise intervention, on cognitive status, physical activity, balance, and biopsychosocial status in people living with PD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with idiopathic Parkinson's disease
* between 1-3 at home according to Modified Hoehn and Yahr Staging (MH&Y)

Exclusion Criteria:

* Individuals who were diagnosed with dementia before Parkinson's diagnosis
* Had undergone deep brain stimulation
* Diagnosed with psychiatric or additional neurological diseases
* Had limited physical activity due to orthopedic problems or previous neurological diseases
* Had communication problems

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire | Three months
  Each question of the BETY-BQ consists of 30 items scored between 0-120 as '0 (never), 1 (yes rarely), 2 (yes sometimes), 3 (yes often), 4 (yes always)'. A high score indicates poor biopsychosocial status.

SECONDARY OUTCOMES:
Beck Depression Scale (BECK-D) | Three months
  It assesses the depression status of individuals. It consists of a total of 21 items assessing unhappiness, self-blame, self-dislike, thoughts of failure, irritability, crying, social withdrawal, indecision, fatigue, insomnia, loss of appetite, somatic distractions, and decreased libido. 1-10: Normal, 11-16: Mild mood changes, 17-20: Borderline clinical depression, 21-30: Moderate depression, 31-40: Severe depression, 40: Very severe depression
International physical activity questionnaire-Short (IPAQ-Short) | Three months
  The scale includes questions about physical activity lasting at least 10 minutes or more in the last 1 week. The IPAQ-Short uses the Metabolic Equivalent (MET) method for physical activity level. Fixed MET values were determined for each section of the scale. These MET values are: Vigorous physical activity, 8 METs; moderate physical activity, 4 METs; walking, 3.3 METs; sitting, 1.5 METs. These MET values are multiplied by the time spent and the number of days, and the results for each activity are summed, and the total MET value is found. Total score values are in MET-minutes/week: Low-level physical activity - Total score < 600 MET min/week, Moderate physical activity - 3000 MET min/week > Total score ≥ 600 MET min/week, High-level physical activity - Total score ≥ 3000 MET min/week.
Berg Balance Scale (BBS) | Three months
  The Berg Balance Scale (BBS) assesses the risk of falling in 14 situations that individuals may encounter daily. Each item is scored between 0-4 in this test according to the individual's ability. While a score of 4 indicates that the individual can complete that item, the highest score can be 56 points.0-20: High fall risk, 21-40: Moderate fall risk, 41-56: Low risk
8-Item Parkinson's Disease Questionnaire (PDQ-8) | Three months
  The 8-item Parkinson's Disease Questionnaire (PDQ-8) consists of one item from each of the eight domains of the PDQ-39 (mobility, activities of daily living, emotional well-being, stigma, communication, social support, cognition, and physical discomfort) with the highest item-total correlation. Each question is scored between 0-4, with a total score in the range of 0-32. A higher score indicates a worse quality of life.
Unified Parkinson's Disease Rating Scale (UPDRS) | Three months
  The scale consists of four parts: 1. Mental, behavioral, and mental status (4 questions), 2. Activities of daily living (13 questions), 3. Motor performance (14 questions), 4. Treatment complications (11 questions). It is used to assess motor impairment and disability in Parkinson's disease. The total score of the scale indicates the severity of the disease. A higher score indicates more severe Parkinson's disease.
Montreal Cognitive Assesment: MoCA | Three months
  The Montreal Cognitive Assessment Test (MoCA) is an assessment tool developed to evaluate mild cognitive impairment. MoCA has items that test executive tasks such as abstract thinking, tracing tests, cube copying, clock drawing, similarity, naming, memory and attention, sentence repetition, verbal fluency, delayed recall, and orientation. This test is scored between 0-30. Cognitive status is considered normal above a total score of 21.
Modified Hoehn & Yahr Staging Scale (MH&Y) | Three months
  It is used to determine the degree of disease and symptoms of Parkinson's disease. The scale has a seven-item staging system.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Alaaddin Keykubat University, Antalya, Alanya
  - Hacettepe University, Ankara, Altındağ

IPD SHARING:
Plan to Share IPD: No
Will not be shared to protect the data of individuals